CLINICAL TRIAL: NCT03653988
Title: Analgesia Efficacy of Pre-operative and Post-operative PEC I/II Block for Bilateral Mastectomy With Reconstruction
Brief Title: Comparison of Pre-op and Post-op Pectoralis Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melinda Seering (Other)
Responsible Party: Sponsor-Investigator, Melinda Seering, Principle Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 201805930
Record Dates: First submitted 2018-08-14; First posted 2018-08-31 (Actual); Results first posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Postoperative Pain; Anesthesia; Nerve Block
Keywords: Nerve block; Pectoralis nerve blocks; PECS I; PECS II; Mastectomy
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CONTROLLED DOUBLE BLIND STUDY
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEC I/II block - pre-operative (Active Comparator): The current standard of care at the University of Iowa is to receive a pectoralis nerve block (PEC I/II) prior to surgery for mastectomy and reconstruction case. The intervention administered to Group I will having the block performed by the anesthesiologist after induction of general anesthesia and prior to surgical incision.
  Interventions: Procedure: PEC I/II blocks by anesthesiologist - pre-operative
- PEC I/II block - intra-operative (Experimental): The current standard of care at the University of Iowa is to receive a pectoralis nerve block (PEC I/II) prior to surgery for mastectomy and reconstruction cases. Group II will have the block administered by the surgeon after mastectomy is performed and before reconstruction.
  Interventions: Procedure: PEC I/II blocks by surgeon - intra-operative

INTERVENTIONS:
Procedure: PEC I/II blocks by anesthesiologist - pre-operative — PEC I/II blocks by anesthesiologist - pre-operative; PEC I/II block to anesthetize the pectoral, intercostobrachial, third to sixth intercostal and long thoracic nerves. The PEC I/II blocks are pectoralis field blocks where local anesthetic medication is injected under ultrasound guidance between the tissue planes of pectoralis major and minor muscles (PECS I) and in the plane of the serratus anterior muscle at the level of the third rib (PEC II). Group I will have the PEC block administered by the anesthesiologist prior to surgical incision.
  Arms: PEC I/II block - pre-operative
Procedure: PEC I/II blocks by surgeon - intra-operative — PEC I/II blocks by surgeon - intra-operative; PEC I/II block to anesthetize the pectoral, intercostobrachial, third to sixth intercostal and long thoracic nerves. The PEC I/II blocks are pectoralis field blocks where local anesthetic medication is injected under ultrasound guidance between the tissue planes of pectoralis major and minor muscles (PECS I) and in the plane of the serratus anterior muscle at the level of the third rib (PEC II).
  Arms: PEC I/II block - intra-operative

SUMMARY:
The investigators will compare whether patients will have better pain control if they were to receive (PEC I/II block) before surgery or after mastectomy.

DETAILED DESCRIPTION:
The current standard of care at the University of Iowa is to receive a pectoralis nerve block (PEC I/II) prior to surgery for mastectomy and reconstruction cases. The investigators will compare whether patients will have better pain control if they were to receive (PEC I/II block) before surgery or after the mastectomy. Patients undergoing mastectomies at the University of Iowa Hospitals clinics receive general anesthesia and a regional block for pain control. The most commonly employed regional anesthetic technique is a PECS I/II block to anesthetize the pectoral, intercostobrachial, third to sixth intercostal and long thoracic nerves. The PECS I/II blocks are pectoralis field blocks where local anesthetic medication is injected under ultrasound guidance between the tissue planes of pectoralis major and minor muscles (PECS I) and in the plane of the serratus anterior muscle at the level of the third rib (PECS II). The investigators will randomize patients into two groups and blind the patient and the research assistant collecting the data. Group I will have the block performed after induction of general anesthesia and prior to surgical incision by the anesthesiologist. Group II will have the block administered by the surgeon after mastectomy is performed and before reconstruction. On the day of surgery, the investigators will have patients fill out forms to measure pain catastrophizing and depression and anxiety. The investigators would like to measure if there is any difference in postoperative pain scores (visual analogue scale)-immediately post surgery in post-anesthesia care unit (PACU), and then on the admission unit every 4 hours for the first twenty four hours or on discharge (whichever time-point occurs sooner) and will collect the average pain scale of the day on post-op day (POD) 2,3,5 and 7 via patient communication electronic message in RedCap. The investigators will also measure intraoperative and post-operative narcotic use (converted to morphine equivalents), post-operative nausea and vomiting, length of (PACU) stay. In addition the investigators will also collect pain scores and pain catastrophic scale on POD 14 after surgery at their clinic visits to the surgeon. Other data collected will include time taken to perform block, post-operative infection rate and post-operative flap necrosis rate.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Female
* Bilateral mastectomy for breast cancer
* Undergoing breast reconstruction
* Must weigh at least 50 kg

Exclusion Criteria:

* More than 80 years of age
* Male
* Prisoners
* Patients who can't provide their own consent
* Lumpectomy only patients
* Patients having prophylactic mastectomies
* Patient must weigh at least 50 kg
* Allergies to local anesthetics
* Patient refusal
* Patients with a history of bleeding disorders
* Non-English speaking patients

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with breast cancer scheduled to undergo mastectomy
Enrollment: 34 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Seering, MD, Principal Investigator — Univerisity of Iowa Hospital & Clinics; Ingrid Lizarraga, MD, Principal Investigator — Univerisity of Iowa Hospital & Clinics
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Access Criteria: IPD will be accessible to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal

REFERENCES:
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] Kamiya Y, Hasegawa M, Yoshida T, Takamatsu M, Koyama Y. Impact of pectoral nerve block on postoperative pain and quality of recovery in patients undergoing breast cancer surgery: A randomised controlled trial. Eur J Anaesthesiol. 2018 Mar;35(3):215-223. doi: 10.1097/EJA.0000000000000762. PMID 29227351
- [Background] Kulhari S, Bharti N, Bala I, Arora S, Singh G. Efficacy of pectoral nerve block versus thoracic paravertebral block for postoperative analgesia after radical mastectomy: a randomized controlled trial. Br J Anaesth. 2016 Sep;117(3):382-6. doi: 10.1093/bja/aew223. PMID 27543533
- [Background] Larsson IM, Ahm Sorensen J, Bille C. The Post-mastectomy Pain Syndrome-A Systematic Review of the Treatment Modalities. Breast J. 2017 May;23(3):338-343. doi: 10.1111/tbj.12739. Epub 2017 Jan 30. PMID 28133848
- [Background] Ruscheweyh R, Viehoff A, Tio J, Pogatzki-Zahn EM. Psychophysical and psychological predictors of acute pain after breast surgery differ in patients with and without pre-existing chronic pain. Pain. 2017 Jun;158(6):1030-1038. doi: 10.1097/j.pain.0000000000000873. PMID 28195858
- [Background] Schreiber KL, Kehlet H, Belfer I, Edwards RR. Predicting, preventing and managing persistent pain after breast cancer surgery: the importance of psychosocial factors. Pain Manag. 2014;4(6):445-59. doi: 10.2217/pmt.14.33. PMID 25494696
- [Background] Schreiber KL, Martel MO, Shnol H, Shaffer JR, Greco C, Viray N, Taylor LN, McLaughlin M, Brufsky A, Ahrendt G, Bovbjerg D, Edwards RR, Belfer I. Persistent pain in postmastectomy patients: comparison of psychophysical, medical, surgical, and psychosocial characteristics between patients with and without pain. Pain. 2013 May;154(5):660-668. doi: 10.1016/j.pain.2012.11.015. Epub 2012 Dec 5. PMID 23290256
- [Background] Vadivelu N, Schreck M, Lopez J, Kodumudi G, Narayan D. Pain after mastectomy and breast reconstruction. Am Surg. 2008 Apr;74(4):285-96. PMID 18453290
- [Background] Vilholm OJ, Cold S, Rasmussen L, Sindrup SH. The postmastectomy pain syndrome: an epidemiological study on the prevalence of chronic pain after surgery for breast cancer. Br J Cancer. 2008 Aug 19;99(4):604-10. doi: 10.1038/sj.bjc.6604534. PMID 18682712
- [Background] Wallace MS, Wallace AM, Lee J, Dobke MK. Pain after breast surgery: a survey of 282 women. Pain. 1996 Aug;66(2-3):195-205. doi: 10.1016/0304-3959(96)03064-3. PMID 8880841
- [Background] Wang L, Guyatt GH, Kennedy SA, Romerosa B, Kwon HY, Kaushal A, Chang Y, Craigie S, de Almeida CPB, Couban RJ, Parascandalo SR, Izhar Z, Reid S, Khan JS, McGillion M, Busse JW. Predictors of persistent pain after breast cancer surgery: a systematic review and meta-analysis of observational studies. CMAJ. 2016 Oct 4;188(14):E352-E361. doi: 10.1503/cmaj.151276. Epub 2016 Jul 11. PMID 27402075
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Kairaluoma PM, Bachmann MS, Rosenberg PH, Pere PJ. Preincisional paravertebral block reduces the prevalence of chronic pain after breast surgery. Anesth Analg. 2006 Sep;103(3):703-8. doi: 10.1213/01.ane.0000230603.92574.4e. PMID 16931684
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Derived] Lizarraga IM, Huang K, Yalamuru B, Mott SL, Sibenaller ZA, Keith JN, Sugg SL, Erdahl LM, Seering M. A Randomized Single-Blinded Study Comparing Preoperative with Post-Mastectomy PECS Block for Post-operative Pain Management in Bilateral Mastectomy with Immediate Reconstruction. Ann Surg Oncol. 2023 Oct;30(10):6010-6021. doi: 10.1245/s10434-023-13890-w. Epub 2023 Aug 1. PMID 37526752

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PEC I/II Block - Pre-operative | PEC I/II Block - Intra-operative
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEC I/II Block - Pre-operative | PEC I/II Block - Intra-operative | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Full Range); unit: years] | 44 [32 to 74] | 44 [44 to 69] | 44 [32 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 17 | 15 | 32
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Assessment Using a Visual Analog Scale-Immediately Post-surgery
Description: The primary outcome to be assessed is to determine if there is a quantitative difference in post-operative pain scores as a result of the administration of a pre-operative PECS I/II block versus the administration of an intra-operative PECS I/II block (Post mastectomy but prior to breast reconstruction). The visual analog scale is a unidimensional measure of pain used in a diverse adult population. The numeric values are on a continuous scale from 0 to 10 with 0 indicating no pain, 5 being moderate pain and 10 as intense pain.
Time Frame: upon arrival to the recovery room after leaving the operating room
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PEC I/II Block - Pre-operative | PEC I/II Block - Intra-operative
Number analyzed (Participants) | 17 | 17
units on a scale | 1.6 [0.3 to 3.0] | 2.3 [1.1 to 3.6]

2. Secondary Outcome: Pain Score Assessment-Post-operative Day 1
Description: Using electronic patient communications, the investigators will ask patients to report their average pain using a numeric values. The numeric values are on a continuous scale from 0 to 10 with 0 indicating no pain, 5 being moderate pain and 10 as intense pain.
Time Frame: Day 1 post surgery
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PEC I/II Block - Pre-operative | PEC I/II Block - Intra-operative
Number analyzed (Participants) | 17 | 17
units on a scale | 3.1 [2.1 to 4.2] | 2.7 [1.6 to 3.7]

3. Secondary Outcome: Pain Score Assessment-Post-operative Day 3
Description: as for outcome 2
Time Frame: Day 3 post surgery
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PEC I/II Block - Pre-operative | PEC I/II Block - Intra-operative
Number analyzed (Participants) | 15 | 16
units on a scale | 2.5 [1.5 to 3.5] | 2.1 [1.0 to 3.1]

4. Secondary Outcome: Pain Score Assessment-Post-operative Day 7
Description: as for outcome 2
Time Frame: Day 7 post surgery
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PEC I/II Block - Pre-operative | PEC I/II Block - Intra-operative
Number analyzed (Participants) | 15 | 16
units on a scale | 1.8 [0.7 to 2.8] | 1.9 [0.8 to 2.9]

5. Secondary Outcome: Pain Score Assessment Using a Visual Analog Scale-Post-operative Surgical Recheck.
Description: When the patient returns to visit with their surgeon approximately 14 days after their surgical procedure, using the visual analog scale the subjects will report their average pain score. The numeric values are on a continuous scale from 0 to 10 with 0 indicating no pain, 5 being moderate pain and 10 as intense pain.
Time Frame: Approximately day 14 post surgery
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | PEC I/II Block - Pre-operative | PEC I/II Block - Intra-operative
Number analyzed (Participants) | 15 | 16
units on a scale | 1.7 [0.6 to 2.7] | 1.2 [0.2 to 2.3]

6. Secondary Outcome: Measure the Amount of Narcotics Use to Control Pain.
Description: The investigators will report the amount of narcotics required (converted to morphine units) to provide pain relief to subjects.
Time Frame: PACU (from time patient left operating room until patient is discharged from the recovery area to in-patient unit). The time limit for this is generally 60-90 minutes
Measure: Median (97.5% Confidence Interval); unit: Morphine Milligram Equivalents
Arm/Group | PEC I/II Block - Pre-operative | PEC I/II Block - Intra-operative
Number analyzed (Participants) | 17 | 17
Morphine Milligram Equivalents | 7.5 [0 to 33] | 8.0 [0 to 40]

7. Secondary Outcome: Measure the Amount of Narcotics Use to Control Pain (In-patient)
Description: as for outcome 6
Time Frame: In-patient (from time patient arrives to in-patient unit from the recovery room until discharged home). Generally this was around 24 hours
Measure: Median (70% Confidence Interval); unit: Morphine Milligram Equivalents
Arm/Group | PEC I/II Block - Pre-operative | PEC I/II Block - Intra-operative
Number analyzed (Participants) | 17 | 17
Morphine Milligram Equivalents | 30 [0 to 75.8] | 25.5 [0 to 90]

8. Secondary Outcome: Measure the Amount of Narcotics Use to Control Pain (Intra-op)
Description: as for outcome 6
Time Frame: Intra-operative (narcotics given during the operating room time)
Measure: Median (99% Confidence Interval); unit: Morphine Milligram Equivalents
Arm/Group | PEC I/II Block - Pre-operative | PEC I/II Block - Intra-operative
Number analyzed (Participants) | 17 | 17
Morphine Milligram Equivalents | 42 [0 to 254] | 42.4 [0 to 108]

ADVERSE EVENTS:
Time Frame: Information collection on adverse events were collected over the first 14 days post-operative
Arm/Group | PEC I/II Block - Pre-operative | PEC I/II Block - Intra-operative
All-Cause Mortality (participants affected / at risk) | 17/17 | 17/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 6/17 | 3/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEC I/II Block - Pre-operative (N=17) | PEC I/II Block - Intra-operative (N=17)
Local Anesthetic Toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEC I/II Block - Pre-operative (N=17) | PEC I/II Block - Intra-operative (N=17)
Vomiting (Surgical and medical procedures) | 6 (6) | 3 (3)

LIMITATIONS AND CAVEATS:
Tools for measuring postoperative pain are subjective. Among the 23 patients who used the electronic reporting format, 58% of the POD 1-14 questionnaires were completed at least one day later, which raises the concern for recall bias. Secondly, our sample size was calculated to detect a difference in mean pain score of 2; however, given the relatively low mean pain scores encountered in our study, this might not be realistic to achieve.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT03653988/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT03653988/SAP_001.pdf
  • Informed Consent Form (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT03653988/ICF_002.pdf